CLINICAL TRIAL: NCT05067205
Title: Minimally Invasive Carpal Tunnel Decompression Using a Novel Ergonomic Releasing Instrument
Brief Title: Minimal Invasive Carpal Tunnel Release With the Novel Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Tien-Ching Lee, Orthopedics Attending Physician, Kaohsiung Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTS001
Record Dates: First submitted 2021-09-08; First posted 2021-10-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open release (Sham Comparator): A prospective, open-label, parallel-group to evaluate the postoperative outcome after carpal tunnel release by using open carpal tunnel release method with duration of 6 months estimated.
  Interventions: Procedure: Carpal tunnel release surgery
- mini CTS releaser (Experimental): A prospective, open-label, parallel-group to evaluate the postoperative outcome after carpal tunnel release by using mini CTS releaser method with duration of 6 months estimated.
  Interventions: Procedure: Carpal tunnel release surgery

INTERVENTIONS:
Procedure: Carpal tunnel release surgery — Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks postoperatively

SUMMARY:
This is a prospective, open-label, parallel-group, randomized controlled trial to evaluate the postoperative outcome after carpal tunnel release by using mini CTS releaser and open method with duration of 6 months estimated.

The study hypothesis is that mini CTS releaser can offer similar functional outcomes to the open approach and avoid the complications of the open surgery.

DETAILED DESCRIPTION:
The current study is the first clinical trial of carpal tunnel syndrome treated by using a device - novel mini CTS releaser. The functional outcome and objective outcome will be recorded to prove the hypothesis that mini CTS releaser can offer similar functional outcomes to the open approach and decrease the complication rate in comparison of the open surgery.

When patients visit, the research physician confirms whether the eligibility criteria are met, and the physician verbally explains the research theme, purpose, and method of execution. After the patient's consent, he should sign the subject consent.

At baseline recruitment, a standardized in-person interview will be conducted by trained and certified study personnel according to structured questionnaires to obtain information on socio-demographic characteristics, habits of tobacco and alcohol use, peripheral blood sample will be also collected from each participant. All of the operated patients underwent a complete personal medical history review, detailed physical examination, as well as routine hematological tests.

Patients will be randomized 1:1 to mini CTS releaser group or to open release group. There will be 35 individuals in each treatment arm. The planned follow-up time will be scheduled.

Safety outcomes including adverse events and changes around surgical wound and neurologic sign will be recorded. Patients will be carefully observed and if any abnormality is noted, appropriate measures will be instituted. The surgical materials used are all certified by the Ministry of Health and Welfare in Taiwan. The possible side effects, such as infections or inflammatory reactions that may occur after surgery, will be given antibiotics or other appropriate treatments in accordance with standard medical procedures.

Data of baseline characteristics will be described using means with standard deviations (SDs) or medians and interquartile ranges (IQRs), or both for continuous variables and using frequencies (percentages) for categorical variables. Mean morphological measures (and changes) will be computed as averages across participants within each treatment group. Between-group baseline comparisons will be based on 2 independent two sample t test or Wilcoxon Mann-Whitney test for quantitative variables, and chi-square test or Fisher's exact test for categorical variables. P values less than 0.05 will be adjusted for multiple comparisons using Bonferroni correction. All statistical analyses will be performed using SAS software Version 9.4 (SAS Institute Inc., Cary, North Carolina).

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age and above.
* clinically symptomatic and electrophysiologically confirmed carpal tunnel syndrome.
* no response to conservative treatment.
* Signed Informed Consent and willing to comply with doctors and nurses' order.

Exclusion Criteria:

* Subjects with recurrent carpal tunnel syndrome
* Subjects with coexisting cervical radiculopathy
* Subjects treated with systemic immunosuppressive or glucocorticosteroids, except subjects taking occasional doses or doses less than 10mg prednisolone per day or equivalent.
* Diabetic patients with pre-OP HbA1c >7%
* Subject included in other ongoing clinical investigation which could interfere with this investigation, as judged by the investigator
* Known allergy/hypersensitivity to any of the components included into the investigation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from preoperative BCTQ SSS at 4 Weeks | preoperative and 4 weeks after surgery
  The Symptom Severity Scale (SSS) of the Boston Carpal Tunnel Questionnaire (BCTQ) is an 11-question patient-administered survey that rates the severity of the patient's carpal tunnel syndrome-specific symptoms on a scale of 1 (no symptoms) to 5 (worst symptoms)

SECONDARY OUTCOMES:
Operation time | operation day
  Outcomes from both interventions will be measured with this symptom severity and functional status carpal tunnel specific scale.
Wound size | Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  Outcomes from both interventions will be measured with this symptom severity and functional status carpal tunnel specific scale.
Grip/pinch strength | Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  Outcomes from both interventions will be measured with this symptom severity and functional status carpal tunnel specific scale.
Pain Scores on the Visual Analog Scale | Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  Is a subjective assessment of pain. The Visual Analogue Scale (VAS) consists of a straight line with the endpoints defining extreme limits such as 'no pain at all' and 'pain as bad as it could be'. The patient is asked to mark his pain level on the line between the two endpoints. The distance between 'no pain at all' and the mark then defines the subject's pain. [0 (no pain), 10 (worst pain)]
Time off work | 24 weeks after surgery
  Differences in time off work between both procedures measured in days.
Number of Participants with Adverse Events | 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  Infection, secondary operation, scar hypertrophy, scar hyper-sensitivity, tenderness, and pillar pain
two point discrimination test | Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  Outcomes from both interventions will be measured with this symptom severity and functional status carpal tunnel specific scale.
BCTQ SSS | Preoperative, 3 days, 2 weeks, 4 weeks and 24 weeks after surgery
  The Symptom Severity Scale (SSS) of the Boston Carpal Tunnel Questionnaire (BCTQ) is an 11-question patient-administered survey that rates the severity of the patient's carpal tunnel syndrome-specific symptoms on a scale of 1 (no symptoms) to 5 (worst symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen HF, Chang SM, Kao CM, Chen YL, Kao LT, Hsu YC, Fu YC, Wang YH, Liu WC, Lee TC. Novel minimally invasive carpal tunnel release using a specialized surgical kit: a prospective multi-center case series. BMC Musculoskelet Disord. 2025 Apr 8;26(1):346. doi: 10.1186/s12891-025-08612-0. PMID 40200263